CLINICAL TRIAL: NCT00238979
Title: A 6-month, 1-arm, Open-label Study to Investigate the Tolerability and Safety of Converting Stable Renal Transplant Recipients Who Receive Tacrolimus With or Without Corticosteroids From Mycophenolate Mofetil (MMF) to Enteric-coated Mycophenolate Sodium (EC-MPS)
Brief Title: A Study to Investigate the Tolerability and Safety of Converting Stable Renal Transplant Recipients Who Receive Tacrolimus With or Without Corticosteroids From Mycophenolate Mofetil (MMF) to Enteric-coated Mycophenolate Sodium (EC-MPS)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CERL080ADE03
Record Dates: First submitted 2005-10-12; First posted 2005-10-14 (Estimated); Last update posted 2011-11-02 (Estimated); Status verified 2011-11

CONDITIONS: Renal Transplantation
Keywords: Renal transplantation, Enteric-coated mycophenolate sodium

INTERVENTIONS:
Drug: Enteric-Coated Mycophenolate Sodium (EC-MPS)

SUMMARY:
The aim of this study is whether a switch of stable renal transplant recipients who receive tacrolimus with or without corticosteroids from mycophenolate mofetil (MMF) to enteric-coated mycophenolate sodium (EC-MPS) is safe and well tolerated by the patients.

ELIGIBILITY:
Inclusion criteria:

* Recipients of first or secondary cadaveric heart-beating, living unrelated or living related kidney transplant.
* Currently receiving 1, 1.5, or 2 g MMF/day, tacrolimus with or without corticosteroids as part of their immunosuppressive regimen for at least 3 months.
* In a stable condition in terms of graft function.

Exclusion criteria:

* Patients who had taken an investigational drug within four weeks prior to study entry
* History of malignancy within the last 5 years, except excised squamous or basal cell carcinoma of the skin.
* Thrombocytopenia (<75,000/mm3), with an absolute neutrophil count of <1,500/mm3 and/or leukocytopenia (<2,500/mm3), and/or hemoglobin <6.0 g/dL prior to enrollment
* Clinically significant infection requiring continued therapy, severe diarrhea, active peptic ulcer disease, or uncontrolled diabetes mellitus, evidence of severe liver disease, HIV or Hepatitis B surface antigen positive.

Other protocol-defined inclusion/exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2003-01; Primary Completion 2005-02 (Actual)

PRIMARY OUTCOMES:
Tolerability based on adverse events within 6 months after switch from MMF to an optimized enteric-coated mycophenolate sodium regimen.

SECONDARY OUTCOMES:
Safety based on renal function within 6 months after medication switch.
Pharmacokinetics of enteric-coated mycophenolate sodium in combination with tacrolimus in a subpopulation at baseline, week 2, month 3
Influence of enteric-coated mycophenolate sodium on the activity of an enzyme at baseline, week 2, month 3
Incidence of biopsy-proven acute rejection, graft loss or death within 6 months post medication switch.
Graft survival and patient survival 6 months post medication switch.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis